CLINICAL TRIAL: NCT05673057
Title: A Phase 1/2a, First-in-human, Open-label, Multicenter, Dose Escalation Study of MP0533 in Patients With Acute Myeloid Leukemia (AML) or Myelodysplastic Syndrome (MDS)
Brief Title: Study of MP0533 in Patients Acute Myeloid Leukemia or Myelodysplastic Syndrome
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Molecular Partners AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MP0533-CP101; 2023-505259-39-00 (EU CTIS Number); 2022-002432-31 (EudraCT Number)
Record Dates: First submitted 2022-12-14; First posted 2023-01-06 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-06

CONDITIONS: Leukemia; Myeloid; Acute; Newly Diagnosed
Keywords: DARPin; CD33; CD123; CD70; T-cell/CD3 engager; multispecific
MeSH Terms: conditions — Leukemia | interventions — Azacitidine; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Dose escalation (Part 1) (Experimental): • MP0533 is administered by intravenous infusion
  Interventions: Drug: MP0533 (multispecific DARPin CD3 Engager Targeting CD33, CD123 and CD70) monotherapy, Part 1
- Dose escalation (Part 2 - Arm A) (Experimental): * MP0533 is administered by intravenous infusion
  * Obinutuzumab pretreatment administered
  Interventions: Drug: MP0533 (multispecific DARPin CD3 Engager Targeting CD33, CD123 and CD70) monotherapy, Part 2-Arm A
- Dose escalation (Part 2 - Arm B) (Experimental): * MP0533 is administered by intravenous infusion
  * Azacitidine is administered by subcutaneous injection for 7 days per cycle
  * Venetoclax is administered orally for 14 days per cycle
  * Optional Obinutuzumab pretreatment administered
  Interventions: Drug: MP0533 (multispecific DARPin CD3 Engager Targeting CD33, CD123 and CD70) + azacitidine + venetoclax
- Dose expansion (Arm A) (Experimental): * MP0533 is administered by intravenous infusion at densified dosing schedule
  * Obinutuzumab pretreatment administered
  Interventions: Drug: MP0533 with Obinutuzumab pretreatment
- Dose expansion (Arm B relapsed/refractory AML) (Experimental): * MP0533 is administered by intravenous infusion
  * Azacitidine is administered by subcutaneous injection for 7 days per cycle
  * Venetoclax is administered orally for 14 days per cycle
  * Optional Obinutuzumab pretreatment administered
  Interventions: Drug: MP0533 + azacitidine + venetoclax with optional Obinutuzumab pretreatment, Arm B in treatment naïve patients
- Dose expansion (Arm B in treatment naïve patients) (Experimental): * MP0533 is administered by intravenous infusion
  * Azacitidine is administered by subcutaneous injection for 7 days per cycle
  * Venetoclax is administered orally for 14 days per cycle
  * Optional obinutuzumab pretreatment administered
  Interventions: Drug: MP0533 + azacitidine + venetoclax with optional Obinutuzumab pretreatment, Arm B relapsed/refractory AML

INTERVENTIONS:
Drug: MP0533 (multispecific DARPin CD3 Engager Targeting CD33, CD123 and CD70) monotherapy, Part 1 — MP0533 is administered by intravenous infusion
  Other Names: Part 1
  Arms: Dose escalation (Part 1)
Drug: MP0533 (multispecific DARPin CD3 Engager Targeting CD33, CD123 and CD70) monotherapy, Part 2-Arm A — * MP0533 is administered by intravenous infusion
  * Obinutuzumab pretreatment administered
  Other Names: Part 2 - Arm A
  Arms: Dose escalation (Part 2 - Arm A)
Drug: MP0533 (multispecific DARPin CD3 Engager Targeting CD33, CD123 and CD70) + azacitidine + venetoclax — * MP0533 is administered by intravenous infusion
  * Azacitidine is administered by subcutaneous injection for 7 days per cycle
  * Venetoclax is administered orally for 14 days per cycle
  * Optional obinutuzumab pretreatment administered
  Other Names: Part 2 - Arm B
  Arms: Dose escalation (Part 2 - Arm B)
Drug: MP0533 with Obinutuzumab pretreatment — * MP0533 is administered by intravenous infusion at densified dosing schedule
  * Obinutuzumab pretreatment administered
  Other Names: Arm A
  Arms: Dose expansion (Arm A)
Drug: MP0533 + azacitidine + venetoclax with optional Obinutuzumab pretreatment, Arm B relapsed/refractory AML — * MP0533 is administered by intravenous infusion
  * Azacitidine is administered by subcutaneous injection for 7 days per cycle
  * Venetoclax is administered orally for 14 days per cycle
  * Optional obinutuzumab pretreatment administered
  Other Names: Arm B relapsed/refractory AML
  Arms: Dose expansion (Arm B in treatment naïve patients)
Drug: MP0533 + azacitidine + venetoclax with optional Obinutuzumab pretreatment, Arm B in treatment naïve patients — * MP0533 is administered by intravenous infusion
  * Azacitidine is administered by subcutaneous injection for 7 days per cycle
  * Venetoclax is administered orally for 14 days per cycle
  * Optional obinutuzumab pretreatment administered
  Other Names: Arm B in treatment naïve patients
  Arms: Dose expansion (Arm B relapsed/refractory AML)

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and preliminary activity of MP0533 in patients with acute myeloid leukemia (AML) or myelodysplastic syndrome (MDS)

ELIGIBILITY:
Inclusion Criteria:

* Has signed and dated written informed consent prior to performing any study procedure, including screening
* Diagnosis of relapsed/refractory AML or relapsed/refractory MDS/AML according to the ELN recommendation 2022.
* Age ≥18 years old on the day of signing informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 to 2
* Anticipated life expectancy ≥ 12 weeks by investigator judgement
* White blood count (WBC) ≤ 15G/L at day of trial drug infusion
* Adequate renal and hepatic function
* Is using highly effective contraception, for females of childbearing potential and for men

Exclusion Criteria:

* Mixed phenotype acute leukemia
* Patients with favorable AML mutations according to ELN recommendation 2022 and 2024
* Allogeneic HCT within the last 3 months and/or eligibility for standard 2nd line of targeted therapy, like gilteritinib for FLT3 mutated AML, unless this therapeutic option has already been given and proven ineffective (patient relapsed or resistant to), or contraindicated, or confounding mutations exist, or there is a lack of access to this recommended therapy.
* More than 2 prior lines of anti-leukemic therapy
* Active GvHD requiring immune-suppressive therapy
* Use of immunosuppressive drugs
* Clinical signs of AML in the central nervous system
* Major surgery within 28 days prior to start of study medication
* Other malignancy requiring active therapy, but adjuvant endocrine therapy is allowed
* Any uncontrolled active infection
* Treatment with investigational agents or agents targeting CD33, CD123 or CD70 within 4 weeks or five times the half-life of the agent, whichever is longer, prior to start of trial medication
* Left ventricular ejection fraction of < 50% on echocardiographic exam at screening
* History or evidence of clinically significant cardiovascular disease
* Pulmonary disease with clinically relevant hypoxia
* Active hepatitis
* Concurrent enrolment in another clinical trial, unless it is an observational (non-interventional) study or it is the follow-up period of an interventional study
* Known hypersensitivity to any of the excipients of the investigational medicinal product (IMP), i.e. finished MP0533 drug

Dose Expansion Group (Arm B in treatment-naïve patients only):

Inclusion

• Treatment-naïve patients who are eligible to AZA+VEN as standard of care

Dose Escalation and Expansion Groups (Arm B only):

Exclusion

1. received VEN in prior treatment lines
2. received strong and/or moderate CYP3A inducers within 7 days before the initiation of AZA/VEN regimen;
3. Has consumed grapefruit, grapefruit products, Seville oranges or Starfruit within 3 days before the initiation of AZA/VEN regimen;
4. Has a malabsorption syndrome or other condition that precludes the enteral route of administration of VEN.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Estimated)
Dates: Start 2022-12-29 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Phase 1 dose escalation: Recommended Phase 2 Dose Regimen and/or Maximum Tolerated Dose Regimen | from start of treatment to end of first cycle (day 1 - 28)
  Incidence of dose limiting toxicities, assessment of toxicity/safety, pharmacokinetic and efficacy parameters
Phase 2 dose extension: Overall Response Rate | throughout the study (on average 3 months)
  Best overall response of complete remission (CR), complete remission with partial hematological recovery (CRh), complete remission with incomplete hematological recovery (CRi), morphologic leukemia-free state (MLFS) and partial remission (PR) according to the European LeukemiaNet (ELN) response criteria 2022

SECONDARY OUTCOMES:
Serum Concentration-time profiles (max. serum) | throughout the study (on average 1 year)
  Determination of PK parameters including (but not limited to) maximum serum concentration (Cmax)
Serum Concentration-time profiles (at Cmax (Tmax)) | throughout the study (on average 1 year)
  Determination of PK parameters including (but not limited to) time at Cmax (Tmax)
Serum Concentration-time profiles (min. serum concentration) | throughout the study (on average 1 year)
  Determination of PK parameters including (but not limited to) minimal serum concentration (Cmin)
Area under the concentration-time curve (AUC) | throughout the study (on average 1 year)
  Pharmacokinetic (PK) analysis of MP0533
Total Clearance (CL) | throughout the study (on average 1 year)
  PK analysis of MP0533
Volume of distribution (Vd) | throughout the study (on average 1 year)
  PK analysis of MP0533
Half-life (t1/2) | throughout the study (on average 1 year)
  PK analysis of MP0533
Incidence of adverse events (AEs) as a measure of safety | throughout the study (on average 1 year)
  Type, incidence and severity of AEs according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0
Event free survival (EFS) | throughout the study (on average 1 year)
  time from the date of first study treatment administration to the date of treatment failure, hematologic relapse from CR/CRh/CRi or death from any cause
Duration of response (DoR) | throughout the study (on average 1 year)
  time from the start date of CR, CRh, CRi, MLFS or PR to relapse or death
Overall survival (OS) | throughout the study (up to 3 years)
  time from the date of first study treatment administration to the date of death
Transfusion-Independence (TI) | throughout the study (on average 1 year)
  portion of subjects who achieved RBC/platelet transfusion independence post baseline
Number of patients proceeding to a stem cell transplantation | throughout the study (on average 1 year)
  Number of patients proceeding to a stem cell transplantation

CONTACTS AND LOCATIONS:
Locations (9):
- France (3):
  - CHU Bordeaux, Bordeaux
  - AP-HP Hôpital Saint-Louis, Paris
  - IUCT Oncopole, Toulouse
- Vilnius University Hospital Santaros Klinikos, Vilnius, Lithuania
- Netherlands (3):
  - Groningen UMC, Groningen, Provincie Groningen
  - Amsterdam UMC - Locatie VUmc, Amsterdam
  - Erasmus MC, Rotterdam
- Switzerland (2):
  - Inselspital, Universitaetsspital Bern, Bern, Canton of Bern
  - Universitaetsspital Zuerich, Zurich, Canton of Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bianchi M, Reichen C, Croset A, Fischer S, Eggenschwiler A, Grubler Y, Marpakwar R, Looser T, Spitzli P, Herzog C, Villemagne D, Schiegg D, Abduli L, Iss C, Neculcea A, Franchini M, Lekishvili T, Ragusa S, Zitt C, Kaufmann Y, Auge A, Hanggi M, Ali W, Frasconi TM, Wullschleger S, Schlegel I, Matzner M, Luthi U, Schlereth B, Dawson KM, Kirkin V, Ochsenbein AF, Grimm S, Reschke N, Riether C, Steiner D, Leupin N, Goubier A. The CD33xCD123xCD70 Multispecific CD3-Engaging DARPin MP0533 Induces Selective T Cell-Mediated Killing of AML Leukemic Stem Cells. Cancer Immunol Res. 2024 Jul 2;12(7):921-943. doi: 10.1158/2326-6066.CIR-23-0692. PMID 38683145